CLINICAL TRIAL: NCT05952258
Title: Magnetic Stimulation as a Treatment for Stress Urinary Incontinence
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Innovation Fund of the Alternative Funding Plan from the Academic Health Sciences Centres of Ontario (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5819
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-07

CONDITIONS: Stress Urinary Incontinence
Keywords: Electromagnetic stimulation therapy
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Double blinded RCT
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnetic stimulation therapy (Active Comparator): Participants will sit fully clothed on the magnetic stimulator chair, with knees apart at about the width of their shoulders, feet flat on the floor. The stimulator will be activated and the intensity gradually increased as tolerated by the participant up to an intensity of 100%. There are a total of 6 treatment sessions (twice per week) over 3 weeks.
  Interventions: Device: Magnetic stimulation
- Sham therapy (Placebo Comparator): Participants will sit fully clothed on the magnetic stimulator chair, with knees apart at about the width of their shoulders, feet flat on the floor. The stimulator will be activated and the intensity gradually increased as tolerated by the participant up to an intensity of 5%. There are a total of 6 treatment sessions (twice per week) over 3 weeks.
  Interventions: Device: Sham Magnetic stimulation

INTERVENTIONS:
Device: Magnetic stimulation — The magnetic stimulation to the pelvic floor muscle will be provided by the Emsella® chair: which will be activated for 28 minutes at each treatment session. The treatment arm will receive up to 100% intensity at each treatment session.
  Arms: Magnetic stimulation therapy
Device: Sham Magnetic stimulation — The sham arm will receive up to 5% intensity at each treatment session
  Arms: Sham therapy

SUMMARY:
The goal of this clinical trial is to determine the efficacy of electromagnetic stimulation treatment of the pelvic floor muscles in adult females with stress urinary incontinence.

DETAILED DESCRIPTION:
A double-blinded randomized controlled clinical trial with a treatment arm and a sham treatment arm will be conducted; followed by an open label trial at 3 months for any sham treatment arm participants who do not meet treatment success.

The primary goal is to compare the subjective success rates for the resolution of stress urinary incontinence (SUI) for the magnetic stimulation treatment at 3 months. Secondary aims include an assessment of complications, resolution of SUI symptoms, patient bother from UI, quality of life and patient satisfaction. The proposed sample size is 158 patients. At the 3-month post treatment evaluation, the treatment allocation will be unmasked. Patients will be followed post treatment up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1) Non-pregnant adult female, not planning pregnancy during the duration of the study 2) Stress urinary incontinence (SUI), as confirmed by history, focused evaluation for ≥3 months 3) objective proof of SUI: Observation of urine leakage by cough and valsalva (positive stress test) at a bladder volume of ≤ 300cc 4) Bladder capacity ≥200cc 5) Post void residual ≤100cc with Stage I or lower pelvic organ prolapse 6) No concurrent or new planned treatment for SUI during the treatment period and the 3 months following it 7) No known body metal from umbilicus to knees 8) Willing and able to comply with the protocol.

Exclusion Criteria:

1) Patient is pregnant, lactating, or plans to become pregnant during the Study; or Patient is <12 months post partum 2) Patient has other predominant type of UI (e.g. Urgency UI, overflow UI, fistula) 3) Current chemo/radiotherapy; history of pelvic radiation; or pelvic surgery < 3 months 4) Systemic diseases known to affect bladder function (e.g. Parkinson's disease, multiple sclerosis, spina bifida, spinal cord injury) 5) Current or history of urethral diverticulum, prior augmentation cystoplasty, implanted nerve stimulators for bladder symptoms 6) Current evaluation or treatment for chronic pelvic pain 7) Participation in another treatment intervention that might interfere with the results of this trial 8) Patient has a medical condition or disorder that may cause non-compliance with the protocol (e.g. unable to perform self-evaluations and/or accurately report medical history, and/or data). 9) Patient has ambulatory 24-hour pad test, where the increased pad weight is < 3 grams. 10) Patient is non-ambulatory (ambulatory with assistive devices allowed) or unable to sit in a chair independently 12) Known body metal located from umbilicus to knees, or cardiac pacemaker 13) Previous magnetic stimulation therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
ICIQ-SF (standardized, validated questionnaire) | 3 months post treatment
  The reporting by the patients of a "cure" at T3 (question #3 of the International Consultation on Incontinence Questionnaire, ICIQ-SF), we have chosen subjective cure as this is the ultimate goal for patients

SECONDARY OUTCOMES:
UDI-6 | 3, 6, 12 and 24 months post treatment
  (standardized, validated questionnaire)
IIQ-7 | 3, 6, 12 and 24 months post treatment
  (standardized, validated questionnaire)
ICIQ-LUTS-qol | 3, 6, 12 and 24 months post treatment
  (standardized, validated questionnaire)
PGI-I | 3, 6, 12 and 24 months post treatment
  (standardized, validated questionnaire)
PISQ-12 | 3, 6, 12 and 24 months post treatment
  (standardized, validated questionnaire)
24 hour pad test | 3 and 12 months
  an objective measure of incontinence and its severity

CONTACTS AND LOCATIONS:
Overall Officials: P Lee, MD, Principal Investigator — Sunnybrook Health Sciences Centre,, University of Toronto
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No